CLINICAL TRIAL: NCT02020954
Title: Prospective Cohort Study of Patients With Mutations in the Dystrophin Gene (X Linked Dilated Cardiomyopathy and Becker Muscular Dystrophy)
Brief Title: Prospective Becker-Heart-Study
Acronym: Becker-HS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Karim WAHBI (Other)
Collaborators: Institut de Myologie, France (Other)
Responsible Party: Sponsor-Investigator, Karim WAHBI, MD, PhD, Institut de Myologie, France
Organization: Institut de Myologie, France (Other)
Other Study IDs: Becker-Heart-Study
Record Dates: First submitted 2013-12-19; First posted 2013-12-25 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Dilated Cardiomyopathy; Lef Ventricular Dysfunction; Heart Failure
MeSH Terms: conditions — Cardiomyopathy, Dilated; Heart Failure | interventions — epicatechin gallate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Dystrophinopathy: Patients with mutations in the DMD gene and Becker muscular dystrophy and/or dilated cardiomyopathy
  Interventions: Procedure: ECG, echocardiography, cardiac MRI, sera biomarkers

INTERVENTIONS:
Procedure: ECG, echocardiography, cardiac MRI, sera biomarkers

SUMMARY:
The purpose of this study is to determine whether electrocardiogram, echocardiography, cardiac MRI, sera biomarkers can improve early detection of myocardial involvement and clinical outcome.

DETAILED DESCRIPTION:
A cohort of 100 patients with mutations in the dystrophin gene associated with Becker muscular dystrophy and/or dilated cardiomyopathy will be included (patients with Duchenne muscular dystrophy are excluded).

Patients with undergo at baseline the following workups: electrocardiogram, echocardiography, cardiac MRI, sera biomarkers measurement.

At 3 years and 5 years, patients will be investigated according to the same protocol and occurrence of cardiac adverse events in the meanwhile will be recorded.

Statistical analysis will assess correlations between cardiac phenotype and DMD mutations and prognostic value of cardiac investigations.

ELIGIBILITY:
Inclusion Criteria:

* mutation in the DMD gene
* Becker muscular dystrophy and/or dilated cardiomyopathy
* age>18 years
* affiliation to the French medical insurance

Exclusion Criteria:

* Duchenne muscular dystrophy
* Any other chronic disease that may be associated with heart disease

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mutations in the DMD gene and Becker muscular dystrophy and/or dilated cardiomyopathy
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Left ventricular ejection fraction | 3 years

SECONDARY OUTCOMES:
Composite endpoint: hospitalisation for heart failure, death due to heart failure | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Karim Wahbi, MD, PhD, Principal Investigator — Institut de Myologie, Cochin Hospital, Paris
Locations (1):
- Institut de Myologie, Paris, Île-de-France Region, France

REFERENCES:
- [Derived] Marty B, Baudin PY, Caldas de Almeida Araujo E, Fromes Y, Wahbi K, Reyngoudt H. Assessment of Extracellular Volume Fraction in Becker Muscular Dystrophy by Using MR Fingerprinting. Radiology. 2023 May;307(3):e221115. doi: 10.1148/radiol.221115. Epub 2023 Mar 7. PMID 36880945